CLINICAL TRIAL: NCT05349916
Title: The Attenuating Effect of Soluble Fiber Consumption on Postprandial Glycemia in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: Grain processing corporation (Unknown)
Responsible Party: Principal Investigator, Bruce R. Hamaker, Distinguished Professor of Food Science, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB-2021-122
Record Dates: First submitted 2021-10-17; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Postprandial Hyperglycemia; Type2 Diabetes; Blood Sugar; High
MeSH Terms: conditions — Hyperglycemia | interventions — isomaltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control (Experimental)
  Interventions: Other: Control
- Isomaltodextrin Low Dose (Experimental)
  Interventions: Other: Isomaltodextrin Low Dose
- Isomaltodextrin High Dose (Experimental)
  Interventions: Other: Isomaltodextrin High Dose
- GPC partially digestible maltodextrin (Experimental)
  Interventions: Other: GPC partially digestible maltodextrin
- Resistant Starch Type 4 (Experimental)
  Interventions: Other: Resistant Starch Type 4

INTERVENTIONS:
Other: Control — 300 g rice porridge + 150 ml drinking water
  Arms: Control
Other: Isomaltodextrin Low Dose — 300 g rice porridge + (5 g IMD in 150 ml drinking water)
  Arms: Isomaltodextrin Low Dose
Other: Isomaltodextrin High Dose — 300 g rice porridge + (10 g IMD in 150 ml drinking water)
  Arms: Isomaltodextrin High Dose
Other: GPC partially digestible maltodextrin — 300 g rice porridge + (15 g GPC fiber in 150 ml drinking water)
  Arms: GPC partially digestible maltodextrin
Other: Resistant Starch Type 4 — 300 g rice porridge + (15 g RS4 starch in 150 ml drinking water)
  Arms: Resistant Starch Type 4

SUMMARY:
The main objective of the current study is to investigate whether consumption of soluble fibers (isomaltodextrin [IMD], partially digestible maltodextrin) and RS4 starch will lower postprandial glycemia as well as postprandial insulin in human subjects with relatively high fasting blood glucose, when consumed with a specific amount of digestible carbohydrate (rice porridge). The primary outcome of the study is the effect of fibers on postprandial blood glucose, whereas the secondary outcome will be its effect on postprandial blood insulin.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (18.5 kg/m² ≤ BMI ≤ 29.9 kg/m²)
* No history of abnormal glucose metabolism
* No ongoing use of drugs affecting blood glucose levels
* Fasting blood glucose between 90-110 mg/dL
* Low dietary fiber intake (less than 15 g per day)

Exclusion Criteria:

* Diabetic individuals
* Individuals with history of gastrointestinal disease
* Pregnant or nursing women

Ages: 22 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2022-03-09 (Actual)

PRIMARY OUTCOMES:
Postprandial glycemic response | Acute study: [3 hours of measurement after consumption of test food]
  Blood glucose will be measured, (AUC)
Postprandial glycemic response | Acute study: [3 hours of measurement after consumption of test food]
  Blood glucose will be measured, (C max)
Postprandial glycemic response | Acute study: [3 hours of measurement after consumption of test food]
  Blood glucose will be measured, (t max)

SECONDARY OUTCOMES:
Postprandial insulin response | Acute study: [3 hours of measurement after consumption of test food]
  Blood insulin will be measured, (AUC)
Postprandial insulin response | Acute study: [3 hours of measurement after consumption of test food]
  Blood insulin will be measured, (C max)
Postprandial insulin response | Acute study: [3 hours of measurement after consumption of test food]
  Blood insulin will be measured, (t max)

CONTACTS AND LOCATIONS:
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: No